CLINICAL TRIAL: NCT01764555
Title: Pharmacokinetics of Intravenous Acetaminophen and Its Metabolites in Morbidly Obese Patients
Brief Title: Pharmacokinetics of Acetaminophen in Morbidly Obese Patients
Acronym: APAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Catherijne Knibbe, Prof. dr., St. Antonius Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APAP study; 2012-000956-32 (EudraCT Number)
Record Dates: First submitted 2012-12-10; First posted 2013-01-09 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal weight patients (Experimental): normal weight patients receiving acetaminophen 2 g instead of 1 g
  Interventions: Drug: acetaminophen 2 g
- mobidly obese patients (Experimental): morbidly obese patients receiving acetaminophen 2 g instead of 1 g
  Interventions: Drug: acetaminophen 2 g

INTERVENTIONS:
Drug: acetaminophen 2 g

SUMMARY:
This study will investigate the pharmacokinetics of acetaminophen in morbidly obese patients versus normal weight patients. Specifically the different metabolic pathways of acetaminophen in morbidly obese adults will be investigated; glucuronidation, sulphation and CYP2E1 (cytochrome P450 2E1) oxidation

ELIGIBILITY:
Inclusion criteria for morbidly obese patients:

* BMI > 40 kg/m2 undergoing bariatric surgery.
* Patients between 18 - 60 years old
* ASA physical classification of II or III
* All racial and ethnic groups will be included

Inclusion criteria for control group:

* BMI between 18 and 25 kg/m2 undergoing general surgery
* Patients between 18 - 60 years old
* ASA (American Society of Anesthesiology) physical classification of I, II or III
* All racial and ethnic groups will be included

Exclusion criteria for all study arms:

* Renal insufficiency
* Liver disease
* Patients with Gilbert-Meulengracht syndrome
* Chronic alcohol intake or use of alcohol within last 72 hours
* Pregnancy or breastfeeding
* Patients who are treated with drugs know to affect CYP2E1 and UGT (UDP glucuronosyltransferase)
* Diabetes mellitus type II patients
* Smoking
* Acetaminophen intake before the study (24 hours before study)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Clearance (total, glucuronidation, sulphation, CYP2E1 oxidation and unchanged) of acetaminophen in morbidly obese patients in comparison with normal weight patients. | 24 hours
Volume of distribution of acetaminophen in morbidly obese patients in comparison with normal weight patients. | 24 hours

SECONDARY OUTCOMES:
Difference in clearance (total, glucuronidation, sulphation, CYP2E1 oxidation) of acetaminophen in morbidly obese patients at the time of bariatric surgery and at 0.5 - 2 year after bariatric surgery. | 8 hours
Difference in volume of distribution of acetaminophen in morbidly obese patients at the time of bariatric surgery and at 0.5 - 2 year after bariatric surgery. | 8 hours
Liver function tests in morbidly obese patients in comparison with normal weight patients. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Catherijne Knibbe, Prof dr, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands